CLINICAL TRIAL: NCT01201772
Title: Impact of Prasugrel Re-load on Platelet Aggregation in Patients on Chronic Prasugrel Therapy
Brief Title: Prasugrel Re-load Strategies
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: UFJ 2010-49
Record Dates: First submitted 2010-09-03; First posted 2010-09-15 (Estimated); Results first posted 2013-01-18 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2011-12

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease; percutaneous coronary revascularization; prasugrel therapy
MeSH Terms: conditions — Coronary Artery Disease | interventions — Prasugrel Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Prasugrel 60mg (Active Comparator): Patients will be randomized to: 10mg, 30mg, or 60mg dose of prasugrel
  Interventions: Drug: Prasugrel
- Prasugrel 30mg (Active Comparator): Patients will be randomized to: 10mg, 30mg, or 60mg dose of prasugrel
  Interventions: Drug: Prasugrel
- Prasugrel 10mg (No Intervention): Patients will be randomized to: 10mg, 30mg, or 60mg dose of prasugrel

INTERVENTIONS:
Drug: Prasugrel — Prasugrel 10mg, 30mg, or 60mg
  Arms: Prasugrel 30mg; Prasugrel 60mg

SUMMARY:
A higher degree of platelet inhibition remains the goal of peri-interventional and long-term anti-thrombotic therapy in patients with coronary artery disease. In clinical practice, patients undergoing percutaneous coronary intervention with stent implantation who are already on clopidogrel therapy get re-loaded with clopidogrel. This is based on prior observations showing that higher inhibition of platelet aggregation may be achieved by giving a loading dose of clopidogrel in patients with coronary artery disease while on chronic clopidogrel therapy. However, to date it is unknown if greater inhibition of platelet aggregation can be achieved by adding a prasugrel loading dose in patients on chronic prasugrel therapy. Therefore, understanding the pharmacodynamic implications of a prasugrel re-load strategy in patients on already on chronic prasugrel therapy will be useful.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with angiographically documented coronary artery disease.
2. Age between 18 to 74 years
3. On treatment with prasugrel 10mg/daily for at least 14 days.

Exclusion Criteria:

1. Blood dyscrasias or bleeding diathesis
2. Antiplatelet treatment with clopidogrel or ticlopidine
3. Recent antiplatelet treatment (< 14 days) with a glycoprotein IIb/IIIa antagonist
4. Platelet count <100x106/µL
5. Active bleeding or hemodynamic instability.
6. Unstable angina, acute or recent (<14 days) myocardial infarction.
7. Serum creatinine >2 mg/dL
8. Baseline ALT >2.5 times the upper limit of normal
9. Oral anticoagulation with a coumarin derivative
10. History of stroke, TIA or intracranial bleeding
11. Weight <60kg
12. Pregnant females

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2010-08; Primary Completion 2011-05 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dominick Angiolillo, MD, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Jacksonville, Florida, United States

REFERENCES:
- [Result] Tello-Montoliu A, Tomasello SD, Ferreiro JL, Ueno M, Seecheran N, Desai B, Kodali M, Charlton RK, Box LC, Zenni MM, Guzman LA, Bass TA, Angiolillo DJ. Pharmacodynamic effects of prasugrel dosing regimens in patients on maintenance prasugrel therapy: results of a prospective randomized study. J Am Coll Cardiol. 2012 May 8;59(19):1681-7. doi: 10.1016/j.jacc.2011.12.039. PMID 22554598

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients recuited at outpatient cardiology clinics
Pre-assignment Details: Seventy-seven patients on maintenance prasugrel therapy were screened. Of these, 11 patients refused to participate in the study and one patient was excluded due to a positive pregnancy test. Thus, a total of 65 patients were randomized.
Groups:
- Prasugrel 10mg: Prasugrel was administered as one 10 mg tablet
- Prasugrel 30mg: Prasugrel was administered as three 10 mg tablet
- Prasugrel 60mg: Prasugrel was administered as six 10 mg tablet
Period: Overall Study
Arm/Group | Prasugrel 10mg | Prasugrel 30mg | Prasugrel 60mg
Started | 23 | 21 | 21
Completed | 22 | 21 | 21
Not Completed | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Prasugrel 30mg: Prasugrel was administered as three 10 mg tablets
- Prasugrel 60mg: Prasugrel was administered as six 10 mg tablets
- Total: Total of all reporting groups
Arm/Group | Prasugrel 10mg | Prasugrel 30mg | Prasugrel 60mg | Total
Number analyzed (Participants) | 23 | 21 | 21 | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 23 | 21 | 21 | 65
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 56 (7) | 54 (7) | 52 (9) | 54 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 3 | 18
  Male | 16 | 13 | 18 | 47
Region of Enrollment [Number; unit: participants]
  United States | 23 | 21 | 21 | 65

OUTCOME MEASURES:

1. Primary Outcome: PRI Levels at 4 Hours
Time Frame: 4 hours after treatment
Population: A total of 65 patients were randomized. One patient assigned to the 10mg prasugrel group was withdrawn after randomization due to anemia identified after baseline blood sampling. Finally, 64 patients [10 mg (n=22), 30 mg (n=21) and 60 mg (n=21)] completed all time periods of the study.
Measure: Mean (Standard Error); unit: percentage of platelet reactivity
Arm/Group | Prasugrel 10mg | Prasugrel 30mg | Prasugrel 60mg
Number analyzed (Participants) | 22 | 21 | 21
percentage of platelet reactivity | 28.8 (2.8) | 11 (2.9) | 2.8 (2.7)

ADVERSE EVENTS:
Groups:
- All Study Participants: All participants who received prasugrel
Arm/Group | All Study Participants
Serious Adverse Events (participants affected / at risk) | 0/65
Other Adverse Events (participants affected / at risk) | 0/65

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No